CLINICAL TRIAL: NCT06836245
Title: Multicenter Application of the Intraoperative Hypothermia Risk Prediction Scale and the Distribution of Risk Factor Characteristics in Surgical Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 016-03-01
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-09

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measure the patient's body temperature intraoperatively using instruments — 1. Core Body Temperature Measurement:
     Nasopharyngeal Temperature Probe: Insert the probe into the patient's nasal cavity to measure the temperature of the nasopharynx.
     Esophageal Probe: Insert the probe through the esophagus to measure the temperature of the lower esophagus.
     Bladder Temperature Probe: Insert the probe into the bladder to measure the temperature of the urine.
     Tympanic Temperature Probe: Place the probe in the ear canal to measure the temperature near the tympanic membrane.
  2. Peripheral Body Temperature Measurement:
  Axillary: Place the thermometer under the armpit, suitable for routine temperature monitoring, but may not be as accurate as core temperature measurement.
  Oral: Place the thermometer under the tongue, suitable for conscious and cooperative patients.
  Rectal: Insert the thermometer into the rectum to provide an accurate temperature measurement, but may not be suitable for all patients, especially those with rectal diseases or immunosuppressed conditions.

SUMMARY:
Research Plan

1.Data Collection and Quality Control

Before the study begins, operating room nursing managers and clinical specialist nurses from 12 participating medical institutions will undergo unified online and offline training on intraoperative hypothermia assessment tools. The training will cover:

1. Risk factor assessment
2. Use of the adult intraoperative hypothermia risk assessment scale
3. Core body temperature measurement
4. Prevention strategies for high-risk patients
5. Management procedures following the occurrence of intraoperative hypothermia After the training, operating room nurses will be assessed on risk factor evaluation and the use of the adult intraoperative hypothermia risk assessment scale to ensure consistency across the 12 institutions. The research team will establish a multi-center database for critically ill surgical patients' intraoperative hypothermia and create a WeChat group for timely communication and problem-solving. Data collection will commence from September to November 2024, lasting three months. Core body temperature measurements will be taken at the following times: upon entering the operating room, baseline core temperature; during surgery, every 30 minutes from skin incision to departure from the operating room. After data collection, all original paper documents will be stored by the researchers, and data will be entered and saved electronically. Both computer data and original documents will be sealed after the study concludes, with all data used solely for this research.

2.Survey Tools

The research data collection tools include:

1. Intraoperative Hypothermia Influencing Factors Collection Form: Collects general information about surgical patients, hypothermia nursing measures, and related influencing factors.
2. Core Body Temperature Record Form: Records the patient's core body temperature from entering to leaving the operating room, with measurements taken every 30 minutes.
3. Adult Intraoperative Hypothermia Risk Assessment Scale: Assessed before surgery by researchers or trained circulating nurses. The study will provide unified definitions and annotations for related hypothermia risk factors to facilitate training and ensure consistency among operating room nurses across the 12 institutions.

3.Data Preservation During the patient's surgery, researchers will use only the pre-designed paper data forms or electronic spreadsheets for data collection, avoiding the use of other electronic devices for activities like photography. The collected patient data will be used exclusively for this study. Patient-related surgical information will not be disclosed to any individuals unrelated to the research, except for sharing with research team members. During statistical analysis, personal privacy information will be removed to minimize the risk of data leakage.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients:

1. Surgical patients aged ≥18 years;
2. The patient or their family members are informed and consent. (Note: The informed consent form requirement for the patient and their family members has been removed from the inclusion criteria. This is because intraoperative hypothermia protection is currently a key aspect of patient surgical care and a major national quality improvement project in medical care. Intraoperative core temperature monitoring and temperature protection measures are required to be routinely performed, and the entire process involves no invasive procedures, so there is no need for a special consent form.)

Exclusion Criteria:

1. Patients undergoing local anesthesia surgery;
2. Surgical patients requiring controlled hypothermic treatment or special intraoperative temperature management;
3. Surgical patients whose underlying disease affects the body's temperature regulation;
4. Patients whose surgical data is incomplete and cannot be collected. (Note: 1. Anesthesia methods are divided into five categories, including local infiltration anesthesia, nerve block anesthesia, epidural anesthesia, non-intubated intravenous general anesthesia, and intubated general anesthesia. Here, surgical patients undergoing local infiltration anesthesia are excluded. 2. Special intraoperative temperature management refers to additional or bundled hypothermia protection measures added to the routine hypothermic care in the operating room.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients from all departments.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Surgical patient body temperature. | 2024.9.15-2025.2.30

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
1. Privacy and Confidentiality: Protecting the privacy of patients is crucial. IPD often contains sensitive personal health information, and unauthorized sharing may violate privacy protection regulations.
  2. Informed Consent: Patients typically need to sign an informed consent form when participating in a study, clearly stating the scope of data usage and sharing. If the consent form does not explicitly authorize sharing of IPD, the data cannot be made public or shared.
  3. Data Security: IPD requires strict security measures to prevent unauthorized access and misuse. Data sharing can only be considered once data security is ensured.
  4. Ethical Guidelines: According to the ethical requirements and approval of the ethics committee, data sharing may be restricted, especially when dealing with vulnerable groups or sensitive diseases.